CLINICAL TRIAL: NCT06298890
Title: Ocular Surface and Corneal Morphological Changes After the Cataract Surgery and Associations With Inflammatory Biomarkers
Brief Title: The Pattern of Dry Eye Disease After Cataract Surgery
Status: Recruiting | Type: Observational
Sponsor: Lithuanian University of Health Sciences (Other)
Collaborators: Santen Oy (Industry)
Responsible Party: Principal Investigator, Reda Zemaitiene, Professor, Head of the Department of Ophthalmology at the Lithuanian University of Health Sciences, Lithuanian University of Health Sciences
Other Study IDs: SASKAT
Record Dates: First submitted 2024-02-22; First posted 2024-03-07 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Dry Eye Disease; Cataract; Ocular Surface Disease
MeSH Terms: conditions — Dry Eye Syndromes; Cataract

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients who will be using artificial tears before and after cataract surgery: Patients will receive artificial tears 7 days before the cataract surgery and continue to use them for 3 months after the surgery.
  Interventions: Device: Artificial tears (sodium hyaluronate 0.2%)
- Patients who will not be using any artificial tears neither before nor after the cataract surgery.: Patients will not receive any artificial tears neither before nor after the cataract surgery.

INTERVENTIONS:
Device: Artificial tears (sodium hyaluronate 0.2%) — Patients randomised into Ist study group will use artificial tears 7 days before the cataract surgery 4 times a day and they will continue to use them after surgery for 3 months.
  Groups: Patients who will be using artificial tears before and after cataract surgery

SUMMARY:
This study is designed to explore dry eye disease (DED) pattern: ocular surface, corneal morphological changes, patients' subjective assessment of DED and their correlations with ocular surface inflammation, pain biomarkers after cataract surgery according to ocular surface lubrication with artificial tears during long-term follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Cataract patients from 50 to 90 years old who underwent uncomplicated phacoemulsification performed by one (and same) experienced surgeon.
* Patients with no underlying ocular surface diseases (keratitis, keratoconjunctivitis and others).
* Patients who previously did not undergo any ophthalmic surgery.

Exclusion Criteria:

* Patient expressed his wish to not participate in the study or discontinue it when already enrolled.
* Severe dry eye disease diagnosed with OSDI/DEQ-5 and at least one of the following tests: TBUT less than 10 seconds, tear osmolarity higher than 308 mOsm/l or positive corneal staining.
* Glaucoma.
* Diabetes mellitus.
* Systemic connective tissue disease, autoimmune disease.
* Neurologic conditions including stroke, Bell's palsy, Parkinson's, trigeminal nerve dysfunction.
* Patients who underwent refractive surgery (LASIK or PRK).
* Contact lens users.
* One or more of the following concomitant medications: psychiatric medicines, antihistamines and/or hormonal replacement.
* Patients who are already regularly using topical drops or ointments.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participation in this study is voluntary. Research participants will be recruited during a routine visit to an ophthalmologist at Lithuanian University of Health Sciences Hospital Kaunas Clinics, Ophthalmology Department.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Assessment of ocular surface changes following cataract surgery | 7 days preoperative, 1 week, 1, 3, 6,12 months postoperative.
  Measured using LacryDiag (Quantel Medical, France), parameters included: non-invasive tear break up time, the height of the tear meniscus, interferometry.
Evaluation of the cornea morphology | 7 days preoperative, 1 week, 1, 3, 6,12 months postoperative.
  Evaluated performing confocal corneal microscopy, parameters include: corneal nerve fibre number and density.
Evaluation of matrix metalloproteinase-9 (MMP-9) levels in patients' tears | 7 days preoperative, 1 week, 1, 3, 6,12 months postoperative.
  Matrix metalloproteinase 9 is an inflammatory biomarker that has been shown to be elevated in the tears of dry eye disease (DED) patients. MMP-9 testing is a valuable diagnostic tool in identifying the presence of ocular surface inflammation in DED patients. MMP-9 level results are classified as positive or negative.
Evaluation of tear osmolarity | 7 days preoperative, 1 week, 1, 3, 6,12 months postoperative.
  Evaluated with the TearLab Osmolarity System. Increased osmolarity indicates dry eye. Values greater than 300 mOsm/kg are suggestive of dry eye. From 300 mOsm/L to 320 mOsm/L, is graded as mild; from 320 mOsm/L to 340 mOsm/L, is graded as moderate; and greater than 340 mOsm/L, is graded as severe.
Evaluation of tear cytokine levels | 7 days preoperative, 1 week, 1, 3, 6,12 months postoperative.
  Interleukin -2, -6, -1β, tumour necrosis factor α (TNFα), interferon-gamma (IFN-γ) levels in tears are significantly higher in patients' with dry eye disease (DED) and they correlate with the severity of DED. Cytokine levels in tears will be evaluated using Human Immunotherapy Luminex® Performance Assay 25-plex Fixed Panel System.
Assessment of central corneal sensitivity | 7 days preoperative, 1 week, 1, 3, 6,12 months postoperative.
  Measured using Cochet-Bonnet aesthesiometer (Luneau; Pruneay-Le-Gillon, France).

SECONDARY OUTCOMES:
Evaluation of potential pain biomarkers in patients' saliva | 7 days preoperative, 1 week, 1, 3, 6,12 months postoperative.
  Pain biomarkers which will be evaluated - soluble tumor necrosis factor-α receptor II (sTNFαRII), nerve growth factor (NGF), brain-derived neurotrophic factor (BDNF), secretory IgA (SIgA). Pain is a common complaint in both dry eye disease (DED) and post-cataract surgery.
  Pain biomarkers will be evaluated using ELISA methods.
Dry Eye Questionnaire-5 (DEQ5) 5-item | 7 days preoperative, 1 week, 1, 3, 6,12 months postoperative.
  The DEQ-5 consists of five questions that assess the following: frequency of watery eye, discomfort, and dryness (scored on a 0-4 scale) and late day discomfort and dryness intensity (scored on a 0 -5 scale).
Ocular surface disease index (OSDI) | 7 days preoperative, 1 week, 1, 3, 6,12 months postoperative.
  OSDI is a 12-item questionnaire that assesses dry eye symptoms and the effects it has on vision-related function in the past week of the patient's life. The questionnaire has 3 subscales: ocular symptoms, vision-related function, and environmental triggers. Patients rate their responses on a 0 to 4 scale with 0 corresponding to "none of the time" and 4 corresponding to "all of the time.
Visual function (VFQ-25) questionnaire | 7 days preoperative, 1 week, 1, 3, 6,12 months postoperative.
  The 25-item questionnaire has several subscale categories that assesses different aspects of health-related quality of life including overall health, overall vision, difficulty with near vision, difficulty with distance vision, limitations in social functioning due to vision, role limitations due to vision, dependency on others due to vision, mental health symptoms due to vision, future expectations for vision, driving difficulties, and pain and discomfort around the eyes
Visual acuity evaluation (LogMAR) | 7 days preoperative, 1 week, 1, 3, 6,12 months postoperative.
  Mean change from baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- Lithuanian University of Health Sciences, Kaunas, Lithuania

IPD SHARING:
Plan to Share IPD: Undecided
If it is necessary (at the motivated request of the customer) to transfer data to the research customer or third parties, only depersonalised data will be transferred, but data transfer to third parties is not foreseen.